CLINICAL TRIAL: NCT02850627
Title: The Effect of Tongguan Capsule for MicroRNA Profiles Between Qi-Stagnation and Qi-Deficiency in Coronary Heart Disease Patients With Blood Stasis Syndrome Undergoing Percutaneous Coronary Intervention
Brief Title: The Effect of Tongguan Capsule for MicroRNA Profiles in Coronary Heart Disease Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Huizheng Zhu, physician, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B2015-129-01
Record Dates: First submitted 2016-07-21; First posted 2016-08-01 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Heart Disease; Acute Myocardial Infarction
Keywords: acute coronary syndrome; Tongguan capsule; miRNAs
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome | interventions — tongguan

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tongguan capsule (Experimental): Tongguan capsule (0.5 g tid. for 6 months)
  Interventions: Drug: Tongguan capsule
- placebo capsule (Placebo Comparator): same volume/day of placebo capsule (0.5 g tid. for 6 months)
  Interventions: Drug: placebo capsule

INTERVENTIONS:
Drug: Tongguan capsule — eligible participants were randomized to receive Tongguan capsule ( 1.5 g/day for six months immediately after PCI)
  Arms: Tongguan capsule
Drug: placebo capsule — eligible participants were randomized to receive placebo capsule ( 1.5 g/day for six months immediately after PCI)
  Arms: placebo capsule

SUMMARY:
The purpose of this study is to test the expression of microRNAs related to the syndromes after the intervention of Tongguan capsule,preliminarily to investigate the mechanism of the effects of Tongguan capsule, and provide the biological foundation of curative effect of Tongguan capsule.

DETAILED DESCRIPTION:
The primary end points is the core of the whole experiment scheme. miRNAs regulate gene expression posttranscriptionally by degrading messenger RNA (mRNA) targets and by blocking their translation Secondary endpoints will include The adverse cardiac clinical events (MACE) in terms of cardiac death,periprocedural myocardial infarction (MI),spontaneous MI and target vessel revascularization(TVR). Related parameters of qi and blood are the material basis of blood conversion and objective performance is used to evaluate the effect on Tongguan capsule on patients with blood stagnation, which can be either interpretation theory of qi deficiency and blood stagnation and mutual transformation between qi and blood can find targets through Tongguan capsule on blood . Routine laboratory tests are used for screening patients basic situation and ensure the safety of the experiment The traditional Chinese medicine syndrome scale Including the the score of deficiency of qi and score of blood stasis syndrome mainly used to identify patients with the traditional Chinese medicine syndrome type Approximately 100 patients in Coronary Heart Disease Patients with Blood Stasis Syndrome undergoing percutaneous coronary intervention will be enrolled and randomized to divided into Qi -stagnation and blood stasis, Qi- deficiency and blood stasis, after the PCI surgery, Qi deficiency and blood stasis group were randomly divided into Tongguan capsule group and the control group, and qi stagnation and blood stasis group, too ,giving patients through Tongguan capsule 3 pills three times a day(1.5g/day), once every three months follow-up, after have been followed up to six months

ELIGIBILITY:
Inclusion Criteria:

1. In line with the diagnostic criteria for acute coronary syndrome (ACS), coronary angiography confirmed for coronary heart disease (CHD), parallel Percutaneous transluminal coronary angioplasty( PTCA) and/or coronary stent implantation was successful
2. Postoperative routine drug treatment
3. Traditional Chinese Medicine syndrome differentiation of qi -deficiency and qi -stagnation blood stasis or blood stasis license
4. Aged 35 to 75 years old
5. Must sign a consent form.

Exclusion Criteria:

1. Renal insufficiency, the male serum creatinine > 2.5 mg/dl (> 220 umo/l), women > 2.0 mg/dl (> 175 umo/l)
2. With obvious liver disease or Alanine aminotransferase ( ALT)， Aspartate aminotransferase ( AST), 3 times higher than normal ceiling
3. Serious cardiac insufficiency (EF < 35%)
4. Uncontrolled patients with high blood pressure
5. Merger or severe valvular heart disease in acute cerebrovascular disease
6. Random blood glucose or greater tendency for 13.7 / L diabetes or glycosylated hemoglobin 9.5% or more
7. Patients with severe mental illness
8. Patients with malignant tumor or life expectancy in less than three years
9. Patients with severe hematopoietic system disease
10. Refused to sign a consent form, or estimated compliance is poorer, follow-up possibilities claim;
11. Pregnancy or ready to pregnant women, nursing mothers;
12. Participated in nearly three months, or is in other clinical subjects . -

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
miRNAs spectrum | six months
  Test the expression of microRNAs related to the syndromes after the intervention of Tongguan capsule,preliminarily to investigate the mechanism of the effects of Tongguan capsule, and provide the biological foundation of curative effect of Tongguan capsule.

SECONDARY OUTCOMES:
major adverse cardiac event | six months
  frequency of the reported cardiovascular events (defined as cardiogenic death, stroke, recurrent myocardial infarction, readmission on account of deterioration of congestive heart failure or unstable angina, target vessel revascularization)
Renin predicts cardiovascular homeostasis and ventricular remodeling | 6 months
  renin（ng/ml） predicts cardiovascular homeostasis and blood pressure maintenance and plays an important role in ventricular remodeling
Ang II predicts cardiovascular homeostasis and ventricular remodeling | 6 months
  Ang II（pg/ml） predicts cardiovascular homeostasis and blood pressure maintenance and plays an important role in ventricular remodeling
Serum E | 6 months
  Acute coronary syndrome is caused by atherosclerotic plaque instability and rupture. The stability of plaque is closely related to inflammation.Serum E (pmol / L) is an important pathway of various immune and inflammatory regulation, which promotes the development of atherosclerosis and is a risk factor for atherosclerosis.
Inflammatory mediators | 6 months
  Tumor Necrosis factor alpha (ng/L)and Interleukin-6，IL-6 (ng/L) measure of the general situation of patients
Brain Natriuretic Peptide | 6 months
  B-type natriuretic peptide（pg/ml） is a neurohormone synthesized in the cardiac ventricles upon ventricular pressure overload and ventricular dilatation
Echocardiography measure of left ventricular systolic function | 6 months
  Evaluation of left ventricular systolic function by left ventricular ejection fraction( LVEF) (%)
Echocardiography measure of left ventricular diastolic function | 6 months
  Left ventricular end diastolic diameter (LVEDD) (mm )measure of left ventricular diastolic function in patients
New York Heart Association functional classification | 6 months
  I Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. no shortness of breath when walking, climbing stairs etc. II Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. III Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest. IV Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Coronary angiography | 6 months
  Quantitative coronary angiography in the stenosis degree, 25%, 50%, 75%, 90%, 99%, 100%, 1, 2, 4, 6, 8,, 16, 32, and, respectively.
  Scoring multiplication will segment coefficients corresponding to the degree of stenosis and the stenosis of total score that is the sum of Gensini score of coronary artery stenosis in the patients.
Seattle Angina Questionnaire score | 6 months
  The Seattle Angina Questionnaire is a valid and reliable instrument that measures five clinically important dimensions of health in patients with coronary artery disease (physical limitation, anginal stability, anginal frequency, treatment satisfaction, and disease perception). (in Units on a Scale).
The traditional Chinese medicine syndrome scale | 6 months
  The traditional Chinese medicine syndrome scale Including the the score of deficiency of qi and score of blood stasis syndrome mainly used to identify patients with traditional Chinese medicine syndrome type

CONTACTS AND LOCATIONS:
Overall Officials: Minzhou Zhang, MD, Study Director — Department of Critical Care Medicine, Guangdong Provincial Hospital of Chinese Medicine; Huizheng Zhu, PhD, Principal Investigator — Department of Critical Care Medicine, Guangdong Provincial Hospital of Chinese Medicine
Locations (1):
- Department of Critical Care Medicine, Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes